CLINICAL TRIAL: NCT01129453
Title: Phase I Trial of a Live Oral Salmonella Enterica Serovar Paratyphi A Vaccine Harboring Mutations in guaBA and clpX
Brief Title: Safety and Immunogenicity of CVD 1902 Oral Attenuated Vaccine to Prevent S. Paratyphi A Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Karen Kotloff, Professor of Pediatrics and Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00045057; Paratyphi CVD 1000 (Other: U. Maryland, Baltimore Center for Vaccine Development); DMID 09-0020 (Other: DMID); U54AI057168 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Salmonella
Keywords: Salmonella; Vaccine
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine-recipients (Experimental)
  Interventions: Biological: CVD 1902, a Salmonella enterica Serovar Paratyphi A live, oral vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CVD 1902, a Salmonella enterica Serovar Paratyphi A live, oral vaccine — CVD 1902 consists of ΔguaBA, ΔclpX Salmonella enterica serovar Paratyphi A vaccine strain diluted in sterile phosphate buffered saline to achieve the desired inoculum. Form: liquid. Dose: 10^6, 10^7, 10^8, or 10^9 CFU per mL. Route: oral.
  Arms: Vaccine-recipients
Other: Placebo — 30 ml of buffer solution (2.0 grams of NaHCO3 dissolved in 150 ml of sterile water) without bacteria, to which food grade corn starch, USP is added, as necessary, to match the turbidity of the vaccine inoculum
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CVD 1902 (a live, attenuated, oral vaccine) is safe and effective in the prevention of Salmonella enterica serovar paratyphi A infection.

DETAILED DESCRIPTION:
Enteric fever is a life-threatening illness caused by several types of a bacterium known as Salmonella, including Salmonella Paratyphi A. In the United States about 400 cases occur each year, and 75% of these are acquired while traveling internationally. Typhoid fever is still common in the developing world, where it affects about 21.5 million persons each year.Besides being a first step towards a possible oral paratyphoid A vaccine for the prevention of enteric fever, this Phase 1 trial will shed light on the suitability of the guaBA,clpX strategy for attenuating non-typhoidal Salmonella, also an emerging pathogens of public health importance. This randomized, double-blinded, Phase I study in healthy is designed to investigate the safety, clinical tolerability, and immunogenicity in a dose escalating fashion of a live, oral, attenuated S. Paratyphi A at four dose levels (10^6, 10^7, 10^8, and 10^9 CFU). We hypothesize that S. Paratyphi A strains harboring mutations in guaBA and clpX will be well tolerated in the full dose range tested and that a single inoculation at the highest dose will elicit vigorous humoral and cell-mediated immune responses in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive
* Good health as determined by a screening evaluation within 35 days before vaccination
* Able to understand and comply with study requirements
* Provides informed, written consent prior to any study procedures
* Agrees to indefinite storage of unused identifiable clinical specimens at the CVD for use in future research, which may require separate IRB approval
* Agrees not to participate in another investigational vaccine or drug trial during the 6-month study; agrees not to receive a licensed vaccine within 14 days of inoculation (if inactivated) or within 30 days of inoculation (if live attenuated)
* If female, has no childbearing potential, i.e., either surgically sterilized or 1 year postmenopausal, or agrees to abstain from becoming pregnant from the day of screening through Day 56 of the trial by using one of the following methods of birth control: abstinence, intrauterine contraceptive device, oral contraceptives or equivalent hormonal contraception (e.g., progestogen-only implantable, cutaneous hormonal patch, injectable contraceptives, or vaginal hormonal ring), diaphragm or condom in combination with spermicide, or is in a relationship with a vasectomized partner
* Agrees not to donate blood to a blood bank for 12 months after receiving the vaccine

Exclusion Criteria:

* An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to:

  * Diabetes mellitus
  * Heart disease (hospitalization for a heart attack or arrhythmia)
  * Seizure disorder (febrile seizures as a child <5 years old or a post-concussive seizure not requiring treatment are acceptable)
  * Recurrent infections (>2 hospitalization for invasive bacterial infections, e.g., pneumonia, meningitis)
  * Immunosuppression as a result of underlying illness or treatment with immunosuppressive drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
  * Active neoplastic disease (or treatment for a neoplastic disease) within past 5 years (excluding non-melanoma skin cancer) or a history of any hematologic malignancy
* Any of the following gastrointestinal conditions:

  • History of any of the following types of abdominal surgery:
* Any major gastrointestinal surgery (e.g., intestinal resection or splenectomy)
* Laparotomy (e.g., hysterectomy, Caesarian section, or appendectomy) within the last 3 years
* Laparoscopic abdominal surgery within the past year

  * A history of cholelithiasis, cholecystitis, other chronic gall bladder disease or empyema of the gall bladder (these subjects can be included only if gall bladder was surgically removed).
  * Crohn's disease, ulcerative colitis, irritable bowel disease, celiac disease, or gastrointestinal ulcers in the past 10 years
  * Bleeding in stool (other than small amounts from straining) in past 12 months
  * Recurrent diarrhea (>5 episodes in past 6 months, each lasting 3 days, with 1 week between them)
* Known allergy or intolerance to penicillins (applicable to women only), ciprofloxacin, trimethoprim/sulfamethoxazole, or corn
* A current illness requiring daily medication other than vitamins, birth control pills, or topical medications
* A history of enteric fever, typhoid fever, or prolonged fever (lasting 3 or more days) within one month after return from international travel, or known exposure to S. Paratyphi or S. Typhi by laboratory work
* A history of having received live oral Ty21a typhoid vaccine or killed whole cell parenteral typhoid vaccine (used by the US Navy into the 1990s)
* Medical, occupational, or family problems resulting from alcohol or illicit drug use in the past 12 months
* Anticipates any of the following during 30 days after discharge from the Inpatient Ward:

  * Shares a household with a child under the age of 3 years
  * Household or sexual contact with someone with weakened immunity (e.g., someone with HIV infection, someone receiving treatment for cancer, a pregnant woman, or an elderly person older than 70 years)
  * Occupation as a foodhandler, childcare (for children <3 years), or health care worker with direct patient contact
* Systolic blood pressure (BP) >150 mm Hg or diastolic BP >90 mm Hg on 2 separate days during medical screening
* A clinically significant abnormality detected on physical examination, including, but not limited to a pathologic heart murmur, lymphadenopathy, hepatosplenomegaly, or a large abdominal scar of unclear origin
* Any of the following laboratory abnormalities detected during medical screening:

  * White blood cell, hemoglobin, or platelet count below the laboratory's lower limit of normal
  * Serum sodium or potassium outside of the laboratory's normal limits
  * Serum creatinine, blood urea nitrogen (BUN), alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (gamma-GTP), bilirubin, prothrombin (PT) or partial thromboplastin time (PTT) above the laboratory's upper limit of normal
  * Fasting glucose >99 mg/dl (if screening >99 mg/dL)
  * Positive serology for hepatitis C or HIV antibody, hepatitis B surface antigen; or syphilis (defined as a positive RPR confirmed by a positive FTA)
  * Stool culture positive for Salmonella, Shigella, Campylobacter, Yersinia, Vibrio cholerae, or lacking normal flora, or pathogenic protozoa by microscopic examination
  * Electrocardiogram (EKG) showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block
* Failure to pass (70% score) a written examination to test for study comprehension
* A woman who is pregnant (positive serum pregnancy test at screening or within 24 h before inoculation) or lactating
* A psychological condition, including a personality, anxiety, or affective disorder, or schizophrenia, which in the opinion of a clinical psychologist compromises the ability of the subject to tolerate the inpatient trial
* Loose stools (Grade 3-5) during the 48-hour acclimatization
* Receipt of any of the following:

  * An investigational vaccine or drug within 30 days of inoculation
  * A licensed vaccine within 14 days (if inactivated) or within 30 days (if live attenuated) of inoculation;
  * Antibiotics within 7 days of vaccination (or within 21 days if the antibiotic was azithromycin);
  * Blood/blood products or immunoglobulins within 6 months prior to the screening visit and/or donation of a unit of blood within 2 months of screening
  * H2 receptor antagonists, proton pump inhibitors, prescription acid suppression medication or over the counter antacids within 72 hours of inoculation
* An oral temperature of 38.3 degrees C (101 degrees F) or higher during the 35-day screening period prior to inoculation
* Other condition(s) that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol
* Poor venous access, defined as the inability to withdraw the required amount of blood for screening tests after 4 attempts

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and clinical acceptability of CVD 1902 with particular attention to febrile adverse reactions and diarrhea during the first 12 days after inoculation, when administered at a dose of either 10^6, 10^7, 10^8, or 10^9 CFU | approximately March 2011
To assess serum antibodies recognizing S. Paratyphi A O polysaccharide and H flagellar antigens, as well as antibody secreting cell (ASC) responses to the O and H antigens as an indication of priming of the mucosal immune system by the vaccine | approximately April 2011

SECONDARY OUTCOMES:
To describe the pattern of fecal shedding of CVD 1902 following vaccination | approximately March 2011
To evaluate the CMI responses, with particular emphasis on antigen-specific cytokine production exhibited by peripheral blood mononuclear cells stimulated with soluble antigens, as well as cytotoxic T lymphocytes to S. Paratyphi-infected autologous cells | approximately March 2011
To evaluate antigen-specific fecal IgA, serum antibodies with functional bactericidal/opsonophagocytic capacity, and magnitude and persistence of memory T and B cell pools as well as functional genomic and proteomic studies | approximately April 2011
To select a well-tolerated and immunogenic dosage level of the vaccine strain for subsequent Phase 2 clinical development | approximately July 2012

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Kotloff, M.D., Principal Investigator — University of Maryland, Baltimore Center for Vaccine Development
Locations (2):
- United States (2):
  - Shin Nippon Biomedical Laboratories (SNBL) Inpatient Facility, Baltimore, Maryland
  - University of Maryland, Baltimore Center for Vaccine Development, Baltimore, Maryland